CLINICAL TRIAL: NCT04828317
Title: Placebo Controlled Alpha-gal Pork Challenge
Brief Title: Alpha-gal Pork Challenge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jeffrey Wilson, MD, Assistant Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: HSR200447
Record Dates: First submitted 2021-03-24; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Allergy;Food
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pork Challenge — Double blind oral challenges comparing wild-type and alpha-gal free pork.

SUMMARY:
This study is investigating the hypothesis that alpha-gal is responsible for the gastrointestinal symptoms that occur in some alpha-gal syndrome subjects following the consumption of mammalian meat. This will be tested by comparing symptoms and immune responses in subjects with alpha-gal syndrome following consumption of "wild-type" pork (which contains alpha-gal) versus consumption of a novel pork product which has been genetically modified to lack alpha-gal (GalSafe pork from Revivicor Inc.).

ELIGIBILITY:
Inclusion Criteria:

Alpha-gal cases:

* Age 18-70
* Patient report of episodic GI symptoms within past 6 months that correlated with ingestion of mammalian meat and/or dairy and which improved on a mammalian avoidance diet.
* IgE to α-Gal >0.1 IU/mL at screening visit.
* Willingness and ability to comply with scheduled visits and study procedures.

Control subjects:

* Age 18-70
* Regularly consume/tolerate mammalian meat without obvious associated gastrointestinal or skin symptoms.
* Have eaten mammalian meat within the past 2 weeks
* Willingness and ability to comply with scheduled visits and study procedures.

Exclusion Criteria:

Alpha-gal cases:

* History of anaphylaxis that was or could have been attributed to mammalian meat in the estimation of the PI.
* IgE to pork which exceeds the value of IgE to α-Gal on screening test
* Unexplained, persistent urticaria or pruritis.
* Pregnancy, breastfeeding or lack of birth control in women of child-bearing age.
* At the discretion of the principal investigator, patients may be excluded due to poorly controlled chronic gastrointestinal conditions including but not limited inflammatory bowel disease (i.e., Crohn's disease, ulcerative colitis, microscopic colitis), acid reflux/heartburn, history of bariatric surgery or gastric banding, active peptic ulcer disease or any abdominal surgery within the past 2 months.
* Patient is unable to swallow food or has poor peripheral access.
* Patient has any medical or physiological disorder or condition that, in the opinion of the Investigator, would compromise the well-being of the patient or study or prevent the patient from meeting or performing study requirements.

Control subjects:

* History of anaphylaxis that was or could have been attributed to mammalian meat in the estimation of the PI
* Unexplained, persistent urticaria or pruritis.
* Poorly controlled chronic gastrointestinal problem
* Patient is unable to swallow food or has poor peripheral access
* Patient has any medical or physiological disorder or condition that, in the opinion of the Investigator, would compromise the well-being of the patient or study or prevent the patient from meeting or performing study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Composite GI symptom score | Score is calculated from survey of gastrointestinal symptoms between 1 and 5 hours after challenge. .
  GI symptoms will be assessed using modified FAST diary. Score is determined from a survey of five gastrointestinal symptoms obtained at 0,1,3,5 hours following oral pork challenge. Symptoms are measured via numerical rating scale (1-5) and aggregate score will be calculated.

SECONDARY OUTCOMES:
Tryptase | Serial samples from 0 to 5 hours post-challenge
  Serum tryptase levels (ng/mL) will be quantified with ImmunoCap comparing post-challenge levels with baseline.
Histamine/Methyl-histamine | Serial samples from 0 to 6 hours post-challenge
  Histamine and methyl-histamine (ng/mL) from serum and urine samples will be quantified with ELISA comparing post-challenge to baseline.
11Beta-PGF2-alpha | Serial samples from 0 to 6 hours post-challenge
  11Beta-PGF2-alpha (pg/mL), a PGD2 metabolite, will be quantified in serum and urine with ELISA comparing post-challenge to baseline

IPD SHARING:
Plan to Share IPD: No